CLINICAL TRIAL: NCT02445690
Title: Correlation Between Thrombin Generation and Endoscopic Activity in Crohn's Disease
Brief Title: Thrombin Generation in Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Other Study IDs: USP
Record Dates: First submitted 2015-05-12; First posted 2015-05-15 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Crohn Disease; Blood Clot; Thrombosis
MeSH Terms: conditions — Crohn Disease; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — 5ml of plasm
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Clinical remission without inflammation: Patients with Crohn's disease in clinical remission and no inflammation in the colonoscopy
- Clinical remission with inflammation: Patients with Crohn's disease in clinical remission and active inflammation in the colonoscopy

SUMMARY:
One hundred and fifty patients with Crohn's disease involving the terminal ileum or the colon, in clinical remission, with or without endoscopic activity will be included. Thrombin generation will be measured and correlated with the simplified endoscopic activity score. The patients will be evaluated for development of deep vein thrombosis after one-year of follow-up.

DETAILED DESCRIPTION:
One hundred and fifty patients with Crohn's disease involving the terminal ileum or the colon, in clinical remission defined by the Crohn's Disease Activity Index below 150 and Harvey-Bradshaw Index below 5, with or without endoscopic activity defined by simplified endoscopic activity score for Crohn's disease (SES-CD) will be included in this study (75 patients with a complete mucosal healing defined by SES-CD below 3 and 75 with endoscopic activity defined by SES-CD above 6) in multiple centers specializing in the treatment of inflammatory bowel diseases in Brazil; Study data will be collected and managed using REDCap electronic data capture tools hosted at the Clinical Hospital of University of São Paulo. REDCap (Research Electronic Data Capture) is a secure, web-based application designed to support data capture for research studies. All thrombin generation tests will be performed at the Clinical Hospital of University of São Paulo, São Paulo, SP through automatically calibrated Thrombogram (CAT- Calibrated Automated Thrombogram®, Maastricht, The Netherlands), with and without thrombomodulin. Those patients will be followed for at least one year after the colonoscopy with measurement of the D-dimer and clinical evaluation every 3 months to verify the developing of deep vein thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Established Crohn's disease diagnosis for at least 6 months
* Disease involvement of the terminal ileum and/or colon
* Clinical remission
* Stable treatment for at least 3 months

Exclusion Criteria:

* Colectomy
* Neoplasia
* Surgery in the last 6 months
* Anticoagulant treatment
* Major liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with established Crohn's disease with stable treatment and clinical remission
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Correlation between thrombin generation and endoscopic activity | At the moment of the inclusion

SECONDARY OUTCOMES:
Association of a high thrombin generation and development of deep vein thrombosis | After 1 year of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Andre ZA Leite, MD, Principal Investigator — Clinical Hospital of São Paulo University
Locations (3):
- Brazil (3):
  - Universidade do Vale do Itajaí-UNIVALI / Santa Catarina, Itajaí, Santa Catarina
  - Faculdade de Medicina de Botucatu -UNESP, Botucatú, São Paulo
  - Clinical Hospital of São Paulo University, São Paulo, São Paulo